CLINICAL TRIAL: NCT04879615
Title: Treatment with Intravenous Alteplase in Ischemic Stroke Patients with Onset Time Between 4.5 and 24 Hours
Brief Title: 24 Hours Treatment with Alteplase in Patients with Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOPE
Record Dates: First submitted 2021-05-06; First posted 2021-05-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alteplase with standard therapy (Experimental)
  Interventions: Drug: Alteplase
- Standard therapy (No Intervention)

INTERVENTIONS:
Drug: Alteplase — Patients will receive standard dose intravenous alteplase (0.9 mg per kilogram, the first 10% administered as an initial bolus and the remainder over a 1-hour period, with a maximum dose of 90 mg)
  Arms: Alteplase with standard therapy

SUMMARY:
The development of intravenous thrombolysis has greatly improved the rate of recanalization and reperfusion in patients with acute ischemic stroke, increasing the proportion of patients with good outcome and reduced mortality. The guideline recommends that patients with ischemic stroke should be treated with intravenous thrombolysis within 4.5 hours. The latest meta-analysis found that ischemic stroke with onset time of 4.5-9 hours with infarction core volume <70ml, ischemic penumbra volume >10ml, and hypoperfusion volume / infarction core volume >1.2 could be benefit from intravenous thrombolysis. The DAWN clinical trial has shown that patients with ischemic stroke with large vessel occlusion with onset time of 6-24 hours could be benefit from endovascular treatment after screening by multi-mode imaging. Therefore, we hypothesize that patients with ischemic stroke with onset time of 4.5-24 hours with a definite penumbra may also benefit from intravenous thrombolysis. The purpose of this study is to explore whether the patients with ischemic stroke with onset time of 4.5-24 hours can benefit from intravenous thrombolysis if they meet the standard of CT perfusion screening.

DETAILED DESCRIPTION:
In recent years, the development of intravenous thrombolysis has greatly improved the rate of recanalization and reperfusion in patients with acute ischemic stroke, increasing the proportion of patients with good outcome and reduced mortality. The guideline recommends that patients with ischemic stroke should be treated with intravenous thrombolysis within 4.5 hours. The latest meta-analysis found that ischemic stroke with onset time of 4.5-9 hours with infarction core volume <70ml, ischemic penumbra volume >10ml, and hypoperfusion volume / infarction core volume >1.2 could be benefit from intravenous thrombolysis (the ratio of mRS 0-1 in 3 months, thrombolysis vs non thrombolysis: 35.4% vs 29.5%). Thus, the time window is not an absolute constant indicator. In theory, compared with time window, the physiological window based on the concept of ischemic penumbra is more reasonable.

In 2015, the AHA/ASA guidelines recommended that patients with ischemic stroke with large vessel occlusion should receive endovascular treatment within 6 hours. The DAWN clinical trial has shown that patients with ischemic stroke with large vessel occlusion with onset time of 6-24 hours could be benefit from endovascular treatment after screening by multi-mode imaging (CT perfusion or MR perfusion). As a result, the 2018 AHA/ASA guidelines extended the endovascular treatment window to 24 hours for patients with large vessel occlusion stroke that meet the standard of perfusion. Therefore, we hypothesize that patients with ischemic stroke with onset time of 4.5-24 hours with a definite penumbra may also benefit from intravenous thrombolysis.

Thus, the purpose of this study is to explore whether the patients with ischemic stroke with onset time of 4.5-24 hours can benefit from intravenous thrombolysis if they meet the standard of CT perfusion screening (infarction core volume <70ml, ischemic penumbra volume >10ml, and hypoperfusion volume / infarction core volume >1.2).

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with clinical signs of acute ischemic stroke between 4.5 and 24 hours from stroke onset, or awakening and unwitnessed stroke (if the midpoint of the last known well time is within 4.5 to 24 hours)
2. Patients aged > 18 years
3. NIHSS range from 4 to 26
4. Imaging inclusion criteria: ischemic core volume ≤ 70 mL, penumbra ≥ 10 mL and mismatch ≥ 20% (as evaluated by CT-perfusion)
5. Pre-stroke mRS score < 2
6. Informed consent has been obtained from the patient, a family member, or a legally responsible person, depending on local ethics requirements

Exclusion Criteria:

1. Intended to proceed to endovascular treatment
2. Contraindications for alteplase:

   * Allergy to alteplase
   * Rapidly improving symptoms at the discretion of the investigator
   * The presence of epileptic seizures, hemiplegia after seizures (Todd's palsy), or other neurological/mental illness that prevents cooperation or willingness to participate
   * Persistent blood pressure elevation (systolic ≥180 mmHg or diastolic ≥100 mmHg) despite treatment
   * Blood glucose levels outside the acceptable range (<2.8 or >22.2 mmol/L, point-of-care glucose testing accepted)
   * High risk of bleeding due to active internal bleeding, major surgery, trauma, gastrointestinal, or urinary tract hemorrhage within the previous 21 days, or arterial puncture at a non-compressible site within the previous 7 days
   * Known impairments in coagulation due to comorbid disease or anticoagulant use, including an INR >1.7 or prothrombin time >15 seconds for those on warfarin, recent use of direct thrombin inhibitors or direct factor Xa inhibitors without reversal capability, or full-dose heparin/heparinoid within the last 24 hours with an aPTT above normal limits
   * Known defect in platelet function or a platelet count below 100,000/mm³
   * History of ischemic stroke, myocardial infarction, intracranial hemorrhage, severe traumatic brain injury, or intraspinal operation within the previous 3 months, or known intracranial neoplasm, arteriovenous malformation, or giant aneurysm
   * Acute or past intracerebral hemorrhage identified by CT or MRI
3. Large (more than one-third of the territory of middle cerebral artery) region of clear hypodensity on CT scan
4. Pregnancy, nursing, or unwillingness to use effective contraceptive measures during the trial period
5. Likelihood of non-adherence to the trial protocol or follow-up
6. Any condition that, in the judgment of the investigator, could impose hazards if study therapy is initiated or affect patient participation in the study
7. Participation in other interventional clinical trials within the previous three months
8. Life expectancy of less than three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Excellent recovery assessed by the ratio of modefied Rankin Scale (mRS) score of 0-1 (%) | at 90 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome

SECONDARY OUTCOMES:
Independent recovery assessed by ratio of modefied Rankin Scale (mRS) score of 0-2 (%) | at 90 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
Ratio of modefied Rankin Scale (mRS) score of 0-3 (%) | at 90 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
Ordinal distribution of mRS score | at 90 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
Major neurologic improvement defined as an improvement of ≥8 points on the NIHSS compared with the initial deficit or a score of ≤1 achieved (%) | at 24 hours
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
Major neurologic improvement defined as an improvement of ≥8 points on the NIHSS compared with the initial deficit or a score of ≤1 achieved (%) | at 7 days
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
Symptomatic intracerebral hemorrhage (sICH) (%) | within 36 hours
  sICH as defined by The European Cooperative Acute Stroke Study III criteria [ECASSIII]
Parenchymal hematoma (PH) (%) | within 36 hours
  PH as defined by the European Cooperative Acute Stroke Study [ECASS] criteria
Mortality (%) | within 90 days
  mortality refers to rate of death from any cause

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Wuwei People's Hospital, Wuwei, Gansu
  - Chongqing University Jiangjin Hospital, Chongqing
  - Binjiang Campus of Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou
  - Bo Ao Campus of Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou
  - Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou
  - Zhejiang Provincial People's Hospital (Affiliated People's Hospital, Hangzhou Medical College), Hangzhou
  - Huzhou Central Hospital, Huzhou
  - First Affiliated Hospital of Jiaxing University, Jiaxing
  - Second Affiliated Hospital of Jiaxing University, Jiaxing
  - The First People's Hospital of Jiashan, Jiaxing
  - The Forth Affiliated Hospital of Zhejiang University, Jinhua
  - Affiliated Hospital of West Anhui Health Vocational College, Liuan
  - Mianyang Hospital of TCM, Mianyang
  - The First People's Hospital of Mianyang (SiChuan Mianyang 404 Hospital), Mianyang
  - Nanjing Lishui District Hospital of Traditional Chinese Medicine, Nanjing
  - Ningbo No. 2 Hospital, Ningbo
  - Zhongshan Hospital, Shanghai
  - Shaoxing People's Hospital (Shaoxing Hospital of Zhejiang University), Shaoxing
  - Suzhou Hospital of Anhui Medical University, Suzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Taizhou First People's Hospital, Taizhou
  - The First People's Hospital of Wenling, Taizhou
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou
  - The People's Hospital of Danyang, Zhenjiang
  - Zhongshan City People's Hospital, Zhongshan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou Y, He Y, Campbell BCV, Liebeskind DS, Yuan C, Chen H, Zhang Y, Yi T, Luo Z, Zhang Z, Meng C, Cheng J, Ouyang H, Hu J, Wang F, Zhang S, Fang Q, Hu H, Zhang X, Chen Y, Zhong W, Lansberg MG, Yan S, Lou M; HOPE investigators. Alteplase for Acute Ischemic Stroke at 4.5 to 24 Hours: The HOPE Randomized Clinical Trial. JAMA. 2025 Sep 2;334(9):788-797. doi: 10.1001/jama.2025.12063. PMID 40773205